CLINICAL TRIAL: NCT03097029
Title: Use of Pancreatic Enzymes in Short Bowel Syndrome
Acronym: SBS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-013255
Record Dates: First submitted 2017-03-24; First posted 2017-03-31 (Actual); Results first posted 2020-03-03 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Short Bowel Syndrome
Keywords: pancreatic enzymes
MeSH Terms: conditions — Short Bowel Syndrome | interventions — Pancrelipase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pancreatic Enzymes (Experimental): All subjects in this study will have exposure to therapy with pancreatic enzymes for a period of about ten days.
  Interventions: Drug: Pancreatic Enzyme

INTERVENTIONS:
Drug: Pancreatic Enzyme — All subjects will take pancreatic enzymes at a dose appropriate for their weight. Pancreatic enzymes are used to help digest fat and other nutrients.
  Other Names: Creon

SUMMARY:
Patients with short bowel syndrome have a high mortality rate that is mainly attributed to complications from central lines and long-term intravenous (IV) nutrition. There are few medical therapies to date that improve gut absorption in patients with short bowel syndrome. The primary objective of this study is to evaluate if absorption from the GI tract improves in subjects with short bowel syndrome following therapy with pancreatic enzymes.

DETAILED DESCRIPTION:
This is an interventional study of subjects with short bowel syndrome to determine if enteral absorption improves following therapy with pancreatic enzymes. The study will assess enteral absorption and nutritional status at baseline through a series of stool tests, blood tests, and anthropometric measurements. Following approximately ten days of therapy with pancreatic enzymes, the study will reassess enteral absorption.

ELIGIBILITY:
Inclusion Criteria:

* history of a small bowel resection with subsequent dependence on parenteral nutrition for at least three months
* age 4 years to 65 years
* usual state of health for the past two weeks with no medication changes
* able to participate in a study for about four weeks with four study visits
* able to take pancreatic enzyme medication orally

Exclusion Criteria:

* significant disease other than short bowel syndrome affecting the gastrointestinal tract that impacts absorption or digestions
* motility disorder
* medications that directly alter fat absorption
* cholestatic liver disease defined as a serum conjugated bilirubin greater than 1.0 mg/dL, chronic renal failure, gout, or hyperuricemia
* history of a pork allergy
* women who are pregnant or lactating
* history of fibrosing colonopathy

Those subjects who are eligible for the malabsorption blood test (MBT) test will be excluded if they have a history of a soy or safflower oil allergy.

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Terry, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sainath NN, Bales C, Brownell JN, Pickett-Blakely O, Sattar A, Stallings VA. Impact of Pancreatic Enzymes on Enteral Fat and Nitrogen Absorption in Short Bowel Syndrome. J Pediatr Gastroenterol Nutr. 2022 Jul 1;75(1):36-41. doi: 10.1097/MPG.0000000000003465. Epub 2022 May 27. PMID 35622082

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pancreatic Enzymes
Started | 15
Completed | 14
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pancreatic Enzymes
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 5
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 10
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Coefficient of Fat Absorption
Description: Coefficient of fat absorption (CFA) measures the amount of fat excreted in the stool compared to how much fat was consumed over the course of 72 hours. This is a measure of fat absorption. CFA was measured at baseline off of pancreatic enzymes and then again while on ten days of pancreatic enzyme supplementation. The change between CFA values at each timepoint was the primary outcome.
Time Frame: Up to 10 days
Population: 3 subjects were not included in the analysis. Two of the subjects did not accurately complete dietary records in order to assess fat intake. One subject submitted such a low stool volume that it was assessed as unlikely to represent a full and accurate stool collection.
Measure: Mean (Standard Deviation); unit: percentage of fat absorbed
Arm/Group | Pancreatic Enzymes
Number analyzed (Participants) | 11
percentage of fat absorbed | 2.3 (13.6)

2. Secondary Outcome: Change in the Coefficient of Nitrogen Absorption
Description: Coefficient of nitrogen absorption (CNA) measures the amount of nitrogen excreted in the stool compared to how much nitrogen was consumed in a 72 hour period. This is a measure of protein absorption. CNA was measured at baseline off of pancreatic enzymes and then again while on ten days of pancreatic enzyme supplementation. The change between CNA values at each timepoint was a study outcome.
Time Frame: Up to 10 days
Population: 3 subjects were not included in the final analysis. Two subjects did not accurately complete a three day dietary record in order to assess nitrogen intake. 1 subject submitted such a low volume of stool that it was assessed as an inaccurate and incomplete stool collection.
Measure: Mean (Standard Deviation); unit: percentage of nitrogen absorbed
Arm/Group | Pancreatic Enzymes
Number analyzed (Participants) | 11
percentage of nitrogen absorbed | 6.9 (15.9)

3. Other Pre Specified Outcome: Change in Malabsorption Blood Test
Description: This test will only be performed on subjects 18 years or older. This an isotope test. Subjects consume a high fat shake with two labeled fats. They have blood tests measured at baseline and then every 1 hour for 8 hours to check for serum levels of labeled fats. This helps determine how well the labeled fats are being absorbed by the intestine.
Time Frame: Up to 10 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data is collected on a daily basis for four weeks, from the time of enrollment (Visit 0), to the final follow-up call (Visit 3). The final study visit was a follow-up telephone call after the subjects were off of the study intervention, pancreatic enzymes. The purpose of this phone call was to assess for adverse events and adherence to the recommended pancreatic enzyme study dose.
Arm/Group | Pancreatic Enzymes
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 8/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pancreatic Enzymes (N=15)
Diarrhea (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Abdominal Pain (Gastrointestinal disorders) | 2
Decreased appetite (Gastrointestinal disorders) | 1
Increased flatus (General disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-06): https://cdn.clinicaltrials.gov/large-docs/29/NCT03097029/Prot_SAP_000.pdf